CLINICAL TRIAL: NCT05606562
Title: Drug-free Without Toothache. A Non-randomized Intervention Study of Free Dental Treatment as a Part of Substance Abuse Treatment.
Brief Title: Drug-free Without Toothache. A Study of Free Dental Treatment as a Part of Substance Abuse Treatment
Acronym: RUST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: #34765
Record Dates: First submitted 2022-02-24; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-02

CONDITIONS: Substance Abuse; Dental Caries
Keywords: Non Randomized Interventional study
MeSH Terms: conditions — Substance-Related Disorders; Dental Caries | interventions — Dental Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental treatment (Experimental): All participants will be offered dental treatment for free.
  Interventions: Procedure: Dental care

INTERVENTIONS:
Procedure: Dental care — Participants will be offered free dental care

SUMMARY:
Objectives: The main objective of the study is to investigate

1. How many patients will attend and complete dental care if they are offered it for free during the stay at "The department of substance abuse treatment, University Hospital North Norway (UNN) in Narvik".
2. Explore whether a parallel dental treatment in addition to the other treatment at the department has a beneficial effect on the abuse treatment, or whether it can be disruptive to offer dental treatment in combination with admission for drug rehabilitation?

DETAILED DESCRIPTION:
This is a non-randomized clinical study without a control group. Approximately 50 persons admitted to "The department of substance abuse treatment (Russeksjon UNN Narvik)" will be offered free dental service during treatment for drug addiction.

ELIGIBILITY:
Inclusion Criteria:

People who are hospitalized for drug abuse at Russeksjon UNN Narvik.

Exclusion Criteria:

Non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dental treatment | Approximately 12 weeks
  Proportion of participant who attend and complete dental treatment during the hospital stay.

SECONDARY OUTCOMES:
Probability measures | Approximately 12 weeks
  Measurement of drop-out from dental treatment. Which factors increase the success of dental treatment (we do not know which factors this will be. This is an exploratory analysis.
Aspects of dental treatment | Approximately 12 weeks
  Will dental treatment have positive or negative impact on drug abuse treatment

CONTACTS AND LOCATIONS:
Overall Officials: Merethe Kumle, MD, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital North Norway, Narvik, Nordland, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT05606562/Prot_000.pdf